CLINICAL TRIAL: NCT07263438
Title: Open-label Phase II Clinical Trial to Test the Efficacy of the Combination of Trimipramine and Atezolizumab With Bevacizumab in Patients With Recurrent Glioblastoma
Brief Title: Efficacy of the Combination of Trimipramine and Atezolizumab With Bevacizumab in Patients With Recurrent Glioblastoma: a Phase 2 Trial
Acronym: Phenix
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Andreas Hottinger, Professor in Neuro-Oncology, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUV- DO-Lundin-PHENIX
Record Dates: First submitted 2025-09-30; First posted 2025-12-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma; Recurrence Tumor
Keywords: recurrent glioblastoma; trimipramine; atezolizumab; bevacizumab
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Trimipramine; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to 2 cohorts based on whether a standard of care surgery is foreseen or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Recurrent GBM without indication for re-resection (Experimental): Eligible patients will receive: trimipramine, bevacizumab and atezolizumab. Trimipramine will be taken orally daily (75 mg the first week and thereafter 150 mg), bevacizumab (15 mg/kg) and atezolizumab (1200 mg) will be administered intravenously every 3 weeks. Maximum treatment duration is 2 years.
  Patients will undergo clinical examination, vital signs measurements, and clinical laboratory evaluations regularly. Safety events will be collected up to 90 days after treatment end.
  Neurological assessment, quality of life assessment, brain Magnetic Resonance Imaging [MRI] and radiological assessment with Response Assessment in Neuro-Oncology [RANO] scale as per local guidelines will be performed every 9 weeks during study treatment administrations. Thereafter, these assessments will be performed every 12 weeks until clinical or radiological recurrence, for up to 3 years after registration.
  Interventions: Drug: Trimipramine; Biological: Cohort 1: Atezolizumab; Biological: Bevacizumab
- Cohort 2: recurrent GBm with an indication for re-resection (Experimental): Eligible patients will receive:
  Trimipramine taken orally daily (75 mg the first week and thereafter 150 mg) and atezolizumab (1200 mg) administered intravenously.
  Neurosurgical resection from first recurrent tumor will be planned 1 cycle after trial treatment start. Trimipramine will be continued during surgery and recovery period (minimum 2 weeks).
  Atezolizumab will be re-started after a minimum recovery period of 14 days after surgery at a fixed dose of 1200 mg administered intravenously, every 3 weeks. Bevacizumab will be started one cycle after the re-start of atezolizumab, at least 35 days after surgery. It will be administered intravenously at a dose of 15 mg/kg every 3 weeks for a maximum of 32 cycles of 21 days.
  Patients will undergo clinical and safety follow-up up to 3 years post-registration as for Cohort 1.
  Interventions: Drug: Trimipramine; Biological: Cohort 2: Atezolizumab; Biological: Cohort 2: Bevacizumab

INTERVENTIONS:
Drug: Trimipramine — Trimipramine: daily oral intake at 75mg/ day for 7 days, then at 150 mg/ day
Biological: Cohort 1: Atezolizumab — Atezolizumab: intravenous administration at 1200 mg on the first day of 3-week cycles.
  Arms: Cohort 1: Recurrent GBM without indication for re-resection
Biological: Bevacizumab — Bevacizumab will be administered intravenously at 15 mg/kg on the first day of 3-week cycles.
  Arms: Cohort 1: Recurrent GBM without indication for re-resection
Biological: Cohort 2: Atezolizumab — Atezolizumab will be administered intravenously at a fixed dose of 1200 mg on the first day of 3-week cycles. Administration will occur once, then will be interrupted during a recovery period of 14-days post surgery, and then resumed.
  Arms: Cohort 2: recurrent GBm with an indication for re-resection
Biological: Cohort 2: Bevacizumab — Bevacizumab will be administered intravenously at 15 mg/kg on the first day of 3-week cycles. The first administration will take place 5 weeks after surgery.
  Arms: Cohort 2: recurrent GBm with an indication for re-resection

SUMMARY:
This is a multicentric phase II open-label clinical trial aiming to assess the efficacy of the combination of trimipramine and atezolizumab with bevacizumab in patients with recurrent glioblastoma. Eligible patients will be assigned to two cohorts depending on whether there is a medical indication for a neurosurgical resection from first recurrent tumor or not.

The aim of the cohort 1 (patients without indication for surgery) is to analyze the clinical efficacy of this triple combination in recurrent glioblastoma. 48 patients will be registered.

The aim of cohort 2 (patients with indication for surgery) is to confirm the level of trimipramine that can be achieved in the tumor tissue and cerebrospinal fluid collected during surgery. At least 5 patients will be registered.

All patients will receive the combination treatment (trimipramine and atezolizumab associated with bevacizumab) for a maximum period of 2 years from registration. The treatment schedule is slightly different for the 2 cohorts because of the neurosurgical resection foreseen for cohort 2 and the requirement to start bevacizumab only after the surgery. After the end of treatment, all patients will be followed up for safety during 90 days from first treatment administration and then up to 3 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed glioblastoma, according to World Health Organization [WHO] 2021 with unequivocal first progression after standard (6 weeks radiotherapy [RT]) with concurrent & adjuvant temozolomide [TMZ] chemotherapy.
* Patients must be at least 3 months off the concomitant part of chemo-radiotherapy.
* Stable or decreasing dose of steroids for 7 days prior to the baseline
* Magnetic Resonance Imaging [MRI] scan.
* Maximum dose of dexamethasone (or equivalent) 4 mg at time of inclusion.
* No surgery or other invasive procedures (major surgical procedure, open biopsy or significant traumatic injury) within 4 weeks prior to registration.
* No core biopsy or other minor surgical procedure within 7 days prior to registration. (Placement of a central vascular access device, if performed at least 2 days prior to trial treatment administration, is allowed).
* Patients who require anti-convulsant therapy must be taking non-enzyme inducing antiepileptic drugs [non-EIAED]. Patients previously on EIAED must be switched to non-EIAED at least 2 weeks prior to registration.
* Measurable disease per Response Assessment in Neuro-Oncology [RANO] version 2.0 criteria. Recurrent disease must be at least one bi-dimensionally measurable contrast-enhancing lesion with clearly defined margins by MRI scan, with minimal diameters of 10 mm, visible on 2 or more axial slices 5 mm apart, based on MRI scan done within 28 days prior to registration.
* Karnofsky performance status 70-100.
* Adequate bone marrow function: neutrophil count ≥ 1.5 x 10^9/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 90 g/L.
* Adequate hepatic function: total bilirubin ≤ 1.5 x Upper Limit of Normal [ULN] (except for patients with Gilbert's syndrome ≤ 3.0 x ULN), aspartate aminotransferase [AST] and alanine transaminase [ALT] and alkaline phosphatase [AP] ≤ 2.5 x ULN.
* Adequate renal function: estimated glomerular filtration rate [eGFR] ≥ 45 mL/min/1.73 m2 (according to Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula).
* Urine dipstick for proteinuria < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hours urine collection and must demonstrate ≤ 1 g of protein/24 hours.
* Adequate coagulation function: International Normalized Ratio [INR] ≤ 1.5 x ULN (the ULN for INR is defined with the value 1.2 for all sites, in case no ULN is documented in the laboratory certificates/sheets). Use of full-dose anticoagulants is permitted as long as the INR is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks before registration, as per American Society for Clinical Oncology [ASCO] guidelines, low molecular weight heparin [LMWH] should be the preferred approach. Concomitant anticoagulation with aspirin (up to 300 mg/day) and anticoagulation with LMWH is allowed.
* Women of childbearing potential must use highly effective contraception , are not pregnant or breast-feeding and agree not to become pregnant during trial treatment and until 6 months after the last dose of investigational drug. A negative pregnancy test before inclusion into the trial is required for all women of childbearing potential.
* Men agree not to donate sperm or to father a child during trial treatment and until 6 months after the last dose of investigational drug.
* Patient is able and willing to swallow trial drug as whole tablet.

Only for Cohort 2:

* Consent to giving access of part of the tumor tissue and Cerebrospinal Fluid [CSF] obtained during the routine neurosurgical procedure for pharmacology and translational studies. Tumor tissue will only be made available once it is established that enough tumor tissue is available for standard neuropathological analysis.
* Patients that have a medical indication for a neurosurgical resection from first recurrent tumor.

Exclusion Criteria:

* Patient must be in first progression/recurrence and have not received more than one line of chemotherapy (concurrent and adjuvant temozolomide). Treatment of Time to Treatment Failure [TTF] fields (Optune®) is allowed during first line but will be stopped at registration.
* Patients must not have prostate enlargement with urinary retention or angle-closure glaucoma at registration.
* Any other experimental drug must be discontinued at least 30 days prior to registration
* Patients under ongoing treatment with an antidepressant must be eligible for a switch to trimipramine. Patients currently under TriCyclic Antidepressant [TCAs] (amitriptyline, clomipramine, nortriptyline, imipramine), selective serotonin reuptake inhibitors (sertraline, paroxetine, fluvoxamine, citalopram, escitalopram) or serotonin and norepinephrine reuptake inhibitors (venlafaxine, duloxetine) must be weaned off these medications for at least 14 days before the introduction of trimipramine.

Note: Patients treated with fluoxetine prior to enrollment will only be eligible for this trial after a two-month washout period before starting the study treatment.

* Prior treatment with atezolizumab or any other immune checkpoint inhibitors.
* Prior treatment with bevacizumab or other Vascular Endothelial Growth Factor [VEGF] inhibitors or VEGF-receptor signaling inhibitors.
* Concomitant or prior use of immunosuppressive medication within 5 half-lives before registration, with the exceptions of intranasal and inhaled corticosteroids.
* Life expectancy of less than 12 weeks.
* Active systemic prior malignancy. Patients with a prior malignancy (basal cell carcinoma of the skin, squamous carcinoma of the skin or carcinoma in situ of the cervix) and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration.
* Blood pressure combination treatment with more than two antihypertensive medications or uncontrolled blood hypertension under properly antihypertensive medications.
* Severe or uncontrolled cardiovascular disease (congestive heart failure New York Heart Association [NYHA] III or IV; unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
* Have a heart rate corrected QT interval using Fridericia's formula [QTcF] (QTc = QT / RR^1/3) ≥ 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g. heart failure, hypokalaemia, familial history of long QT interval syndrome). Patients with bundle branch block and prolonged QTcF are permitted with approval of the sponsor investigator.
* Presence of a grade 3 atrioventricular [AV] block on electrocardiogram [ECG].
* History of cerebrovascular accident or intracranial haemorrhage within 6 months prior to registration.
* Known history of human immunodeficiency virus [HIV] or active chronic hepatitis C or hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous antimicrobial treatment.
* Known history of tuberculosis, known history of primary immunodeficiency, known history of allogeneic organ transplant. Receipt of live attenuated vaccine within 28 days prior to the first dose of atezolizumab administration. Vaccination with inactivated viruses, such as those in the influenza vaccine, are permitted.
* History of or active auto-immune disease with the exception of diabetes mellitus type II and well controlled hypothyroidism on treatment.
* Concomitant treatment with strong or moderate cytochrome P450 3A or 2D6 [CYP3A or CYP2D6] inducers or inhibitors.
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information.
* Monoamine oxidase inhibitors [MAOI] (Rasagiline, or others not approved in Switzerland, such as phenelzine, tranylcypromine, isocarboxazid and selegiline). Of note, MAOI must have been stopped at least 14 days prior to the start of trimipramine.
* Known hypersensitivity to trial drug(s) or to any component of the trial drug(s)
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Progression-free survival rate [PFSR] | 6 months after last patient's registration
  Progression-free survival rate [PFSR]: evaluated at 6 months after registration using the Response Assessment in Neuro-Oncology [RANO] verion 2.0 critieria
Cohort 2: Level of trimipramine in the tumor tissue and cerebrospinal fluid [CSF] | 3 months after last patient's surgery
  Level of trimipramine in the tumor tissue and CSF collected during surgery will be assessed by measuring the trimipramine concentration by laboratory analysis.

CONTACTS AND LOCATIONS:
Locations (6):
- Switzerland (6):
  - Universitätsspital Basel, Basel, Basel
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Bern Inselspital, Bern, Canton of Bern
  - Luzerner Kantonsspital, Lucerne, Canton of Lucerne
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Universitätsspital Zürich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Undecided